CLINICAL TRIAL: NCT00960427
Title: Colorectal Cancer Stem Cells Marker Expression in Rectal Cancer Patients Undergoing Chemoradiotherapy-A Pilot Study
Brief Title: Studying Biomarkers in Tumor Tissue and Blood Samples From Patients Undergoing Chemotherapy and Radiation Therapy for Stage II or Stage III Rectal Cancer That Can Be Removed By Surgery
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: No surgeon available to perfrom gastroscopy
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000649658; WSU-2009-041 (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2009-08-14; First posted 2009-08-17 (Estimated); Last update posted 2013-04-16 (Estimated); Status verified 2013-04

CONDITIONS: Colorectal Cancer
Keywords: adenocarcinoma of the rectum; stage II rectal cancer; stage III rectal cancer
MeSH Terms: conditions — Colorectal Neoplasms; Rectal Neoplasms | interventions — Neoadjuvant Therapy; Gene Expression Profiling; Reverse Transcriptase Polymerase Chain Reaction; Immunohistochemistry; Endoscopic Mucosal Resection; Sigmoidoscopy; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: systemic chemotherapy
Genetic: RNA analysis
Genetic: gene expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: immunohistochemistry staining method
Other: laboratory biomarker analysis
Procedure: endoscopic biopsy
Procedure: neoadjuvant therapy
Procedure: sigmoidoscopy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Studying samples of tumor tissue and blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This phase I trial is studying biomarkers in tumor tissue and blood samples from patients undergoing chemotherapy and radiation therapy for stage II or stage III rectal cancer that can be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To obtain the distribution of stem cell markers (CD166, CD44, and ESA) in tumor tissue samples before and after neoadjuvant chemoradiotherapy (NCRT) in patients with stage II or III rectal cancer.

Secondary

* To correlate disease-free survival after NCRT with baseline expression and change in expression of stem cell markers (CD166, CD44, and ESA) after NCRT.
* To correlate baseline and post-NCRT expression of all three stem cell markers (CD166, CD44, and ESA) with circulating tumor cell (CTC) count and stem cell marker expression on CTC at baseline and after NCRT.

OUTLINE: Patients receive chemotherapy according to the treating physician's choice and undergo concurrent radiotherapy over approximately 6 weeks. Between 6-8 weeks after completion of neoadjuvant chemoradiotherapy (NCRT), patients undergo low anterior or abdominoperineal surgical resection. Some patients may then receive additional chemotherapy.

Tumor tissue samples are obtained via sigmoidoscopy-guided biopsies at baseline and at the time of surgery. Blood samples are also collected at baseline and after completion of NCRT. Samples are isolated for RNA analysis of CD44, CD166, and ESA expression by quantitative reverse transcriptase-PCR and IHC.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed adenocarcinoma of the rectum

  * Inferior margin within 16 cm of the anal verge on endoscopic exams
* Locally advanced or low lying disease meeting 1 of the following stage criteria:

  * Stage II (T2, N0, M0) disease

    * Distal tumor (< 5 cm from anal verge) invades into muscularis propria but not beyond (T2)
  * Stage II (T3-4, N0, M0) disease

    * Tumor invades through muscularis propria into subserosa or into non-peritonealized pericolic or perirectal tissues (T3) OR tumor directly invades other organs or structures and/or perforates visceral peritoneum (T4)
  * Stage III (any T, N1-2, M0) disease

    * Tumor has invaded to any depth with involvement of regional lymph nodes (N1-2)
* Resectable disease
* No suspicious metastatic disease (M1)

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* Adequate organ function
* No significant co-morbidities that would preclude the use of neoadjuvant chemoradiotherapy, including any of the following:

  * Severe heart failure
  * Arrhythmia
  * Significant liver or kidney dysfunction
* No psychiatric or addictive disorder that would preclude study compliance
* No bleeding diathesis
* No contraindication for sigmoidoscopy

PRIOR CONCURRENT THERAPY:

* No prior radiotherapy or chemotherapy for rectal cancer
* No concurrent warfarin unless appropriate bridging therapy is arranged during biopsy procedures

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Estimation of stem cell markers with stated precision
Correlation of disease-free survival with post-treatment value and change in expression of colorectal cancer stem cell markers after neoadjuvant chemoradiotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Bhaumik B. Patel, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute